CLINICAL TRIAL: NCT02663063
Title: The Application of Evidence-Based Chinese Complementary and Alternative Medicine (CAM) in Hospice Palliative Care in Taiwan-The Second and Third Year Project.
Brief Title: CAM in Hospice Palliative Care in Taiwan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2015-10-005A
Record Dates: First submitted 2016-01-21; First posted 2016-01-26 (Estimated); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Cancer
Keywords: Complementary and alternative medicine; Hospice Palliative Care
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SSP treatment group (Experimental): Case on SSP treatment
  Interventions: Device: SSP treatment
- Non-SSP treatment group (Sham Comparator): Sham SSP treatment
  Interventions: Device: SSP treatment

INTERVENTIONS:
Device: SSP treatment — SSP treatment 5 times a week

SUMMARY:
The study aims to explore the effects of silver spike point (SSP) treatment on common symptoms including pain, breathlessness, nausea/vomiting, dry mouth etc. of terminal cancer patients.

DETAILED DESCRIPTION:
The study aims to explore the effects of silver spike point treatment on common symptoms including pain, breathlessness, nausea/vomiting, dry mouth etc. of terminal cancer patients. We will conducted a pilot study to evaluate the effects on different symptoms and then a prospective study will be conducted after validation of major effects.

ELIGIBILITY:
Inclusion Criteria:

* Cancer patients
* Competent with clear consciousness
* With symptoms of pain, breathlessness, nause/vomiting, dry mouth, generalized discomfort
* Expected life span of at least 1 week

Exclusion Criteria:

* With implanted devices
* Not having clear consciousness
* Expected life span less than 1 week
* Foreigner

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-12; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Symptom severity score | One week after treatment
  Questionnaire for evaluating the severity of symptoms

SECONDARY OUTCOMES:
Quality of life | One week after treatment
  Questionnaire for evaluating quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Shinn-Jang Hwang, MD, Principal Investigator — Taipei Veterans General Hospital, Taipei, Taiwan
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
Undecided

REFERENCES:
- [Background] Bausewein C, Booth S, Gysels M, Higginson I. Non-pharmacological interventions for breathlessness in advanced stages of malignant and non-malignant diseases. Cochrane Database Syst Rev. 2008 Apr 16;(2):CD005623. doi: 10.1002/14651858.CD005623.pub2. PMID 18425927
- [Background] Chen FP, Chen TJ, Kung YY, Chen YC, Chou LF, Chen FJ, Hwang SJ. Use frequency of traditional Chinese medicine in Taiwan. BMC Health Serv Res. 2007 Feb 23;7:26. doi: 10.1186/1472-6963-7-26. PMID 17319950
- [Background] Chiu TY, Hu WY, Chen CY. Prevalence and severity of symptoms in terminal cancer patients: a study in Taiwan. Support Care Cancer. 2000 Jul;8(4):311-3. doi: 10.1007/s005209900112. PMID 10923772
- [Background] Deng G, Hou BL, Holodny AI, Cassileth BR. Functional magnetic resonance imaging (fMRI) changes and saliva production associated with acupuncture at LI-2 acupuncture point: a randomized controlled study. BMC Complement Altern Med. 2008 Jul 7;8:37. doi: 10.1186/1472-6882-8-37. PMID 18606019
- [Background] Enblom A, Johnsson A, Hammar M, Onelov E, Steineck G, Borjeson S. Acupuncture compared with placebo acupuncture in radiotherapy-induced nausea--a randomized controlled study. Ann Oncol. 2012 May;23(5):1353-1361. doi: 10.1093/annonc/mdr402. Epub 2011 Sep 23. PMID 21948812
- [Background] Enblom A, Lekander M, Hammar M, Johnsson A, Onelov E, Ingvar M, Steineck G, Borjeson S. Getting the grip on nonspecific treatment effects: emesis in patients randomized to acupuncture or sham compared to patients receiving standard care. PLoS One. 2011 Mar 23;6(3):e14766. doi: 10.1371/journal.pone.0014766. PMID 21448267
- [Background] Ernst E, Lee MS. Acupuncture for palliative and supportive cancer care: a systematic review of systematic reviews. J Pain Symptom Manage. 2010 Jul;40(1):e3-5. doi: 10.1016/j.jpainsymman.2010.03.010. No abstract available. PMID 20619198
- [Background] Garcia MK, Chiang JS, Cohen L, Liu M, Palmer JL, Rosenthal DI, Wei Q, Tung S, Wang C, Rahlfs T, Chambers MS. Acupuncture for radiation-induced xerostomia in patients with cancer: a pilot study. Head Neck. 2009 Oct;31(10):1360-8. doi: 10.1002/hed.21110. PMID 19378325
- [Background] Garcia MK, McQuade J, Haddad R, Patel S, Lee R, Yang P, Palmer JL, Cohen L. Systematic review of acupuncture in cancer care: a synthesis of the evidence. J Clin Oncol. 2013 Mar 1;31(7):952-60. doi: 10.1200/JCO.2012.43.5818. Epub 2013 Jan 22. PMID 23341529
- [Background] Hervik J, Mjaland O. Quality of life of breast cancer patients medicated with anti-estrogens, 2 years after acupuncture treatment: a qualitative study. Int J Womens Health. 2010 Sep 28;2:319-25. doi: 10.2147/IJWH.S12809. PMID 21151679
- [Background] Jedel E. Acupuncture in xerostomia--a systematic review. J Oral Rehabil. 2005 Jun;32(6):392-6. doi: 10.1111/j.1365-2842.2005.01445.x. PMID 15899016
- [Background] Lang DS. Nonpharmacologic interventions for breathlessness in advanced stages of malignant and nonmalignant diseases. Clin J Oncol Nurs. 2012 Jun 1;16(3):320. doi: 10.1188/12.CJON.320. No abstract available. PMID 22641326
- [Background] Lewis CR, de Vedia A, Reuer B, Schwan R, Tourin C. Integrating complementary and alternative medicine (CAM) into standard hospice and palliative care. Am J Hosp Palliat Care. 2003 May-Jun;20(3):221-8. doi: 10.1177/104990910302000312. PMID 12785044
- [Background] Meng Z, Kay Garcia M, Hu C, Chiang J, Chambers M, Rosenthal DI, Peng H, Wu C, Zhao Q, Zhao G, Liu L, Spelman A, Lynn Palmer J, Wei Q, Cohen L. Sham-controlled, randomised, feasibility trial of acupuncture for prevention of radiation-induced xerostomia among patients with nasopharyngeal carcinoma. Eur J Cancer. 2012 Jul;48(11):1692-9. doi: 10.1016/j.ejca.2011.12.030. Epub 2012 Jan 28. PMID 22285177
- [Background] O'Sullivan EM, Higginson IJ. Clinical effectiveness and safety of acupuncture in the treatment of irradiation-induced xerostomia in patients with head and neck cancer: a systematic review. Acupunct Med. 2010 Dec;28(4):191-9. doi: 10.1136/aim.2010.002733. Epub 2010 Nov 9. PMID 21062848
- [Background] Standish LJ, Kozak L, Congdon S. Acupuncture is underutilized in hospice and palliative medicine. Am J Hosp Palliat Care. 2008 Aug-Sep;25(4):298-308. doi: 10.1177/1049909108315916. Epub 2008 Jun 6. PMID 18539767
- [Background] Sugimoto K, Konda T, Shimahara M, Hyodo M, Kitade T. A clinical study on SSP (silver spike point) electro-therapy combined with splint therapy for temporo-mandibular joint dysfunction. Acupunct Electrother Res. 1995 Jan-Mar;20(1):7-13. doi: 10.3727/036012995816357177. PMID 7572330
- [Background] Tseng KL, Liu HJ, Tso KY, Woung LC, Su YC, Lin JG. A clinical study of acupuncture and SSP (silver spike point) electro-therapy for dry eye syndrome. Am J Chin Med. 2006;34(2):197-206. doi: 10.1142/S0192415X0600376X. PMID 16552832
- [Background] Vickers AJ, Cronin AM, Maschino AC, Lewith G, MacPherson H, Foster NE, Sherman KJ, Witt CM, Linde K; Acupuncture Trialists' Collaboration. Acupuncture for chronic pain: individual patient data meta-analysis. Arch Intern Med. 2012 Oct 22;172(19):1444-53. doi: 10.1001/archinternmed.2012.3654. PMID 22965186
- [Background] Vickers AJ, Cronin AM, Maschino AC, Lewith G, Macpherson H, Victor N, Sherman KJ, Witt C, Linde K; Acupuncture Trialists' Collaboration. Individual patient data meta-analysis of acupuncture for chronic pain: protocol of the Acupuncture Trialists' Collaboration. Trials. 2010 Sep 28;11:90. doi: 10.1186/1745-6215-11-90. PMID 20920180
- [Background] Wong R, Sagar CM, Sagar SM. Integration of Chinese medicine into supportive cancer care: a modern role for an ancient tradition. Cancer Treat Rev. 2001 Aug;27(4):235-46. doi: 10.1053/ctrv.2001.0227. PMID 11545543
- [Background] Xu W, Towers AD, Li P, Collet JP. Traditional Chinese medicine in cancer care: perspectives and experiences of patients and professionals in China. Eur J Cancer Care (Engl). 2006 Sep;15(4):397-403. doi: 10.1111/j.1365-2354.2006.00685.x. PMID 16968323
- [Background] Zhuang L, Yang Z, Zeng X, Zhua X, Chen Z, Liu L, Meng Z. The preventive and therapeutic effect of acupuncture for radiation-induced xerostomia in patients with head and neck cancer: a systematic review. Integr Cancer Ther. 2013 May;12(3):197-205. doi: 10.1177/1534735412451321. Epub 2012 Jul 12. PMID 22791311